CLINICAL TRIAL: NCT01582295
Title: Dose Finding Pilot Study of Cabozantinib (XL184) Administered Orally as Monotherapy for the Treatment of Patients With Relapsed or Relapsed/Refractory Multiple Myeloma With Bone Disease
Brief Title: XL184 For Relapsed/Refractory Multiple Myeloma (MM) With Bone Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-005
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Bone disease
MeSH Terms: conditions — Multiple Myeloma; Bone Diseases | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Cabozantinib ( XL 184)
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Starting dose 40 mg daily
  Other Names: XL 184

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational drug. Phase I studies also try to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. It also means the FDA has not approved the drug for your type of cancer.

Cabozantanib (XL184) is a new drug that is being developed to treat cancer. The study drug cabozantinib works by inhibiting several different proteins which are believed to be involved in multiple myeloma growth, its ability to spread, and its ability to form new blood vessels. This drug has been used in other research studies and information from those other research studies suggests that this drug may help to slow or stop disease growth to bones and prevent cancer growth.

In this research study, we are looking to see how effective cabozantanib is in slowing or stopping disease growth to the bones as well as preventing your cancer from worsening. We are also looking for the highest dose of cabozantinib that can be given safely to patients who have multiple myeloma with bone disease.

DETAILED DESCRIPTION:
Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have multiple myeloma, not everyone who participates in this research study will receive the same dose of study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

The study drug, cabozantinib, comes in the form of tablets which you will take by mouth. You will take your dose of cabozantinib once a day during each 28 day cycle.

Detailed instructions on how to take the study drug and which foods and drinks you will be prohibited from taking during the research study can be found in your study drug diary.

During Cycle 1, you will come into the clinic weekly (Day 1, 8, 15 and 22). For all other cycles, you will come into the clinic on Day 1 and 15.

A visit will be scheduled 30 days after you have finished or stopped taking the study drug so your doctor will be able to check your well being.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/Refractory Multiple Myeloma
* Skeletal lesions suggestive of bone involvement
* Must have received at least 2 lines of prior systemic therapy for the treatment of multiple myeloma
* Must have received prior treatment with a proteasome inhibitor
* Agree to use medically accepted barrier method of contraception
* Not a candidate for ASCT, has declined the option or has relapsed after prior ASCT

Exclusion Criteria:

* Pregnant or breastfeeding
* Has received radiotherapy to thoracic cavity or GI tract (within 3 months of first dose of study drug), bone or brain metastasis (within 14 days of first dose) or any other site (within 28 days)
* Has received any other investigational agent within 28 days
* Primary brain tumor
* Uncontrolled, significant intercurrent or recent illness
* Cardiovascular disorder(s)
* Gastrointestinal disorder(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety of Cabozantinib | 2 years
  To determine the safety of cabozantinib in patients with multiple myeloma with bone disease

SECONDARY OUTCOMES:
Changes in Biochemical Markers | 2 years
  Changes in biochemical markers of bone turnover, including serum bone specific alkaline phosphatase, osteocalcin, sclerostin, P1nP (procollagen type 1N propeptide) and urine N-telopeptide before treatment and end of cycle 2
Effect of Cabozantinib on Bone Disease | 2 years
  To evaluate the effect of cabozantinib on bone disease as assessed by post-treatment changes on whole body FDG-PET/CT scan before treatment and end of cycle 2
Objective Response per IMWG | 2 years
  Objective response according to the International Myeloma Working Group Uniform Response Criteria (IMWG)
Pain Assessment | 2 years
  Pain will be assessed using the Pain Assessment Tool included in the appendix. The questionnaire will be administered at screening, day 1 of each cycle and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Yee, MD, Principal Investigator — Massachusetts General Hospital, Boston
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts